CLINICAL TRIAL: NCT04696289
Title: Predicting Pediatric Intraluminal Pulmonary Vein Stenosis Outcomes Using a Comprehensive Standardized Catheterization Assessment
Brief Title: Predicting Pediatric Pulmonary Vein Stenosis Outcomes Using Data Acquired During a Cardiac Catheterization
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Ryan Callahan, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-P00035534
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Vein Stenosis
MeSH Terms: conditions — Stenosis, Pulmonary Vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized catheterization assessment (Experimental): Assessment of pulmonary veins including angiography, intravascular ultrasound, pressure assessment and compliance testing.
  Interventions: Diagnostic Test: Standardized catheterization assessment

INTERVENTIONS:
Diagnostic Test: Standardized catheterization assessment — There are four components to the pulmonary vein assessment.
  1. Angiography: pulmonary artery wedge injection and/or selective pulmonary vein injection.
  2. Intravascular ultrasound: manual pullback of IVUS catheter from lobar segment to left atrium.
  3. Pressure assessment: pulmonary vein pressure (mmHg) measured before and after (if applicable) intervention.
  4. Compliance testing: the compliance of the vein will be measured using a compliant conventional balloon.

SUMMARY:
This is a prospective, single center study which applies a standardized, comprehensive catheterization assessment to patients with a known or suspected diagnosis of pulmonary vein stenosis (PVS) who are undergoing a cardiac catheterization at Boston Children's Hospital. As part of the assessment, each pulmonary vein will undergo angiography (pictures using moving x-rays and contrast dye), intravascular ultrasound (IVUS; pictures of the vein wall using a catheter inside the vein), pressure assessment and compliance testing. The status of each pulmonary vein will then be assessed 12 months after the catheterization (i.e. no disease, severe disease, etc.). Using statistics, the investigators will determine which patient and vein characteristics (obtained at the of catheterization) can predict whether or not a pulmonary vein will have disease. The investigators hypothesize that this comprehensive, standardized, invasive assessment of pediatric intraluminal PVS can predict vein outcome.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing cardiac catheterization for the indication of known or suspicion for intraluminal pulmonary vein stenosis.

Exclusion Criteria:

* Hemodynamically unstable patients as determined by the patient care team.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vein status | 12 months +/- 6 weeks or prior to study exit due to death or lung transplant
  Severity of pulmonary vein stenosis (score 0 to 3); Score 0: Unobstructed vein (best outcome), Score 1: Proximal vein disease, Score 2: Distal vein disease, Score 3: Vein atresia (worst outcome).

SECONDARY OUTCOMES:
Patient status | 12 months
  Transplant free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Esch, MD, Principal Investigator — Boston Children's Hospital/Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadr IM, Tan PE, Kieran MW, Jenkins KJ. Mechanism of pulmonary vein stenosis in infants with normally connected veins. Am J Cardiol. 2000 Sep 1;86(5):577-9, A10. doi: 10.1016/s0002-9149(00)01022-5. PMID 11009286
- [Background] Kovach AE, Magcalas PM, Ireland C, McEnany K, Oliveira AM, Kieran MW, Baird CW, Jenkins K, Vargas SO. Paucicellular Fibrointimal Proliferation Characterizes Pediatric Pulmonary Vein Stenosis: Clinicopathologic Analysis of 213 Samples From 97 Patients. Am J Surg Pathol. 2017 Sep;41(9):1198-1204. doi: 10.1097/PAS.0000000000000892. PMID 28622179
- [Background] Callahan R, Kieran MW, Baird CW, Colan SD, Gauvreau K, Ireland CM, Marshall AC, Sena LM, Vargas SO, Jenkins KJ. Adjunct Targeted Biologic Inhibition Agents to Treat Aggressive Multivessel Intraluminal Pediatric Pulmonary Vein Stenosis. J Pediatr. 2018 Jul;198:29-35.e5. doi: 10.1016/j.jpeds.2018.01.029. Epub 2018 Mar 23. PMID 29576325
- [Background] Callahan R, Jenkins KJ, Gauthier Z, Gauvreau K, Porras D. Preliminary findings on the use of intravascular ultrasound in the assessment of pediatric pulmonary vein stenosis. Catheter Cardiovasc Interv. 2021 Feb 15;97(3):E362-E370. doi: 10.1002/ccd.29264. Epub 2020 Sep 16. PMID 32936535
- [Derived] Callahan R, Gauvreau K, Keochakian M, Esch JJ, Porras D, Bergersen L, Beroukhim R, Farias M, Harrild DM, Ireland CM, Kwatra N, Jenkins KJ. Predicting Outcomes in Pediatric Intraluminal Pulmonary Vein Stenosis Using a Comprehensive Standardized Catheterization Assessment: A Prospective Study. Circ Cardiovasc Interv. 2025 Sep;18(9):e015002. doi: 10.1161/CIRCINTERVENTIONS.124.015002. Epub 2025 Jul 14. PMID 40654078